CLINICAL TRIAL: NCT04096677
Title: Effects of Hysteroscopy and Transvaginal Surgery on Reproductive Prognosis and Endometrium Receptive in Patients With Post Cesarean Scar Defect
Brief Title: Effects of Hysteroscopy and Transvaginal Surgery on Reproductive Prognosis in Patients With Post Cesarean Scar Defect
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yuqing Chen, Deputy chief physician, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: Post cesarean scar defect
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Post Cesarean Scar Defect; Hysteroscopy
Keywords: post cesarean scar defect; hysteroscopy; transvaginal intervention; endometrial receptive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — endometrium
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hysteroscopy repair: patients with post cesarean scar defect
  Interventions: Procedure: hysteroscpy
- transvaginal repair: patients with post cesarean scar defect

INTERVENTIONS:
Procedure: hysteroscpy
  Groups: hysteroscopy repair

SUMMARY:
The study is to compare hysteroscopic repair and transvaginal intervention for correcting uterine defect in patients with post cesarean scar defect (PCSD) and the reproductive prognosis.

DETAILED DESCRIPTION:
Post cesarean scar defect (PCSD), refers the lower uterine segment form a reservoir-like pouch during healing process after transverse lower uterine segment cesarean section connected with uterine cavity. The pouch has a valve-like effect, obstructing blood drainage and accumulating blood in depression. These causes may lead to a variety of gynecological disturbances, secondary dysmenorrheal and infertility. Some patients can occur some serious obstetric complications, such as cesarean scar pregnancy and even the rupture of uterus during a subsequent pregnancy. At present, the causes and mechanisms of PCSD are not clear, diagnosis and treatment are not uniform. Surgical methods include abdominal surgery, laparoscopic surgery, transvaginal surgery, hysteroscopic surgery, hysteroscopic with laparoscopic surgery and so on. Hysteroscopic and transvaginal surgery to treating PCSD both are minimally invasive and feasible surgical approach. However, hysteroscopic surgery and transvaginal surgery have not been compared for correcting the uterine defect in patients with PCSD before.

ELIGIBILITY:
Inclusion Criteria:

* Patients had a history of transverse lower uterine segment cesarean section;
* Patients had a previous regular menstruation, while after caesarean section, they occurred prolonged postmentrual bleeding (10-20days)
* Medication failed(contraceptive pills).
* Sex hormone test is normal;
* TVU or hysteroscopy showed a triangular or U-shaped anechoic liquid dark area and on the anterior lower uterine segment in relation to cesarean section scar during menstruation of 7-12 days or hysteroscopic examination showed uterine anterior wall defect like dome changes at isthmus below internal orifice of cervix.

Exclusion Criteria:

* Irregular menstrual cycle before cesarean section
* Previous placement of an intrauterine contraceptive device
* Presence of other organic uterine pathology responsible for abnormal uterine bleeding, such as endometrial hyperplasia, polyps or submucosal myomas, cervical cancer, endometrial cancer, etc
* Existence of endocrine diseases, such as dysfunction of pituitary, ovarian, adrenal gland, and thyroid;
* Coagulation dysfunction.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients who received hysteroscopy in the Department of Obstetrics and Gynecology of the First Affiliated Hospital of Sun Yat-sen University and were diagnosed with post cesarean scar defect according to the transvaginal ultrasonography or hysteroscopy were recruited into present study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a less postoperative menstruation | 6 months
  Follow-up carried out 6 months after the initial operation, using the following criteria to evaluate curative effect: Cure: menstrual duration was shortened to no more than 7 days and TVU showed no liquid dark area in scar of lower uterine segment; Improvement: menstrual duration was reduced by more than 2 days, but menstrual duration was still longer than 7days and TVU showed the liquid dark area in lower segment of uterus disappeared or narrowed. Failure: menstrual duration was reduced by less than 2 days or had no obvious change, and TVU showed the liquid dark area in lower segment of uterus did not narrow. Efficiency rate = cure rate + improvement rate.
Number of Participants being a pregnant | 1 year
  Follow-up carried out 1 year after the initial operation, postoperative pregnancy with a history of infertility preoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Yuqing Chen, Study Chair — The First Affiliated Hospital of SunYetSen University
Locations (2):
- China (2):
  - First affiliated hospital of SUN Yat-Sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of SunYetSen University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Yes